CLINICAL TRIAL: NCT03179293
Title: Transition to Propofol After Sevoflurane Anaesthesia to Prevent Emergence Agitation in Genito-urinary Paediatric Surgeries
Brief Title: Transition to Propofol After Sevoflurane Anaesthesia to Prevent Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: propofol after sevo
Record Dates: First submitted 2017-06-03; First posted 2017-06-07 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol (Active Comparator): propofol 1 mg/kg IV bolus will be given to the patient with a further 2 mg/kg administered manually over the next 3 min prior to the patient leaving the OR
  Interventions: Drug: Propofol
- Control (Placebo Comparator): Normal saline will be administered IV over the next 3 min prior to the patient leaving the OR
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Propofol — propofol 1 mg/kg IV bolus will be given to the patient with a further 2 mg/kg administered manually over the next 3 min prior to the patient leaving the OR
  Arms: Propofol
Drug: Normal saline — Normal saline will be administered manually over the next 3 min prior to the patient leaving the OR
  Arms: Control

SUMMARY:
The aim of this randomized double-blinded study is to determine whether transition to propofol for 3 min at the end of sevoﬂurane anaesthesia reduces the incidence of EA in children undergoing genito-urinary paediatric surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Children Aged 3 - 8 years
2. ASA (I - II)
3. Genito-urinary Surgeries: hernia, varicocele, etc.

Exclusion Criteria:

1. Patients or parental refusal
2. Allergy to Propofol or egg products; or a family history of malignant hyperthermia
3. Operating time more than 60 minutes
4. Performance of any other procedure under the same anaesthetic
5. Presence of co-morbidities or congenital anomalies
6. mental disease, neurologic disease, treatment with sedatives, full stomach, or indication for rapid sequence induction.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Emergence Agitation | 30 min after emergence
  The incidence of EA according to the Watcha scale (deﬁned as a score ≥3 at any time in the 30 min after emergence)
Emergence Agitation | 30 min after emergence
  The incidence of EA according to the Paediatric Emergence Anaesthesia Delirium (PAED) scale (deﬁned as a score >12 at any time in the 30 min after emergence )

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No